CLINICAL TRIAL: NCT03027362
Title: Cognitive Therapy to Sustain the Antidepressant Effects of Intravenous Ketamine in Treatment-resistant Depression: a Randomized Controlled Trial
Brief Title: Cognitive Therapy to Sustain the Antidepressant Effects of Intravenous Ketamine in Treatment-resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1609018450
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (CBT) and medication (Experimental): Following clinical ketamine treatment, the intervention includes sixteen CBT sessions over 14 weeks. In addition, standard of care medications for treatment of depression, will be prescribed by the principal investigator or by a psychiatrist unaffiliated with the trial. Participants will remain on the medication they were prescribed when they entered the study and will be expected not to adjust the medication unless clinically urgent.
  Interventions: Other: Cognitive behavioral therapy (CBT) and medication
- Psychoeducation and medication (Active Comparator): Following clinical ketamine treatment, the intervention includes psychoeducational sessions over 14 weeks.In addition, standard of care medications for treatment of depression, will be prescribed by the principal investigator or a by psychiatrist unaffiliated with the trial.
  Interventions: Other: Psychoeducation and medication

INTERVENTIONS:
Other: Cognitive behavioral therapy (CBT) and medication — Sixteen sessions over 14 weeks.
  Arms: Cognitive behavioral therapy (CBT) and medication
Other: Psychoeducation and medication
  Arms: Psychoeducation and medication

SUMMARY:
The goals of this study are: 1) to investigate the efficacy of combining ketamine with intensive cognitive behavioral therapy (CBT) to sustain the antidepressant effects of ketamine; and 2) to determine ketamine's delayed effects on learning and memory, and to explore the relationship between any ketamine-induced changes in learning and memory and duration of antidepressant efficacy, with and without CBT augmentation. Subjects with a diagnosis of MDD who are treatment-resistant to at least 2 antidepressants and have chosen to pursue clinical ketamine treatment at Yale Psychiatric Hospital will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a major depressive episode based on Diagnostic and Statistical manual (DSM) 5 criteria and having failed one or more standard antidepressant treatments during the current episode
* Hamilton Depression Rating Scale (17-HAM-D) score of 21 or more prior to ketamine treatment.
* Planned clinical treatment with ketamine at Yale Psychiatric Hospital (YPH)
* As the purpose of this study is to determine the feasibility and efficacy of CBT to sustain the antidepressant effects of ketamine, only those who achieve a clinical response (i.e., 50% reduction in depression symptoms, as measured by the Montgomery-Asberg Depressive Rating Scale (MADRS) will be eligible for randomization.
* Patients must be treatment resistant to at least two drugs used to treat depression.

Exclusion Criteria:

* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their depressive episode or has been predominant to their depressive episode at any time within 6 months prior to screening
* Active suicidal thoughts with a plan
* Current or recent (<6 months ago) substance use disorder
* Non-affective psychosis (such as schizophrenia or schizoaffective disorder)
* Inability to speak English fluently
* A clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results
* Dementia, delirium, or any other neurological or mental disease that might affect cognition or the ability to meaningfully participate in cognitive behavioral therapy (CBT).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Time to relapse of depression measured by the Montgomery-Asberg Depressive Rating Scale (MADRS) score. | Enrollment to 17 week follow-up
  Relapse is defined as less than 50% improvement in MADRS compared to baseline MADRS score. The median time to relapse is the time at which the 50th percentile of participants relapses.

SECONDARY OUTCOMES:
Change in cognitive flexibility-working memory | Before the first ketamine treatment and 24 hours following the last ketamine treatment.
  Measured by n-back task
Change in cognitive flexibility-executive function | Before the first ketamine treatment and 24 hours following the last ketamine treatment.
  Measured by set shifting task (COGSTATE test)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wilkinson, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States